CLINICAL TRIAL: NCT00515762
Title: Pilot Trial of Prevention of Persistent Alopecia Following Docetaxel by Means of Scalp Cooling (ELASTO-GEL CAPS)in Breast Cancer Patients
Brief Title: Prevention of Persistent Alopecia Following Docetaxel by Means of Scalp Cooling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Miguel Martin, MD, Hospital San Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALOPER-2
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-06

CONDITIONS: Alopecia; Breast Cancer
Keywords: persistent alopecia; docetaxel; breast cancer
MeSH Terms: conditions — Alopecia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1: scalp cooling (Experimental): scalp cooling
  Interventions: Device: elasto-gel cap

INTERVENTIONS:
Device: elasto-gel cap — scalp cooling cap

SUMMARY:
Persistent alopecia following adjuvant docetaxel for breast cancer is a side-effect that has been recently described. This pilot trial explores the capacity of a cooling cap (Elasto-gel) to prevent persistent alopecia in breast cancer patients treated with adjuvant docetaxel regimens.

DETAILED DESCRIPTION:
Persistent alopecia following adjuvant docetaxel for breast cancer is a side-effect that has been recently described. Docetaxel is toxic to skin and skin annexes and can produce nail toxicity and persistent alopecia. Nail toxicity has been successfully prevented by means of hypothermic gloves and slippers (Elasto-gel, Southwest Technologies, Inc, North Kansas City, MO). This pilot trial explores the capacity of a cooling cap (Elasto-gel) to prevent persistent alopecia in breast cancer patients treated with adjuvant docetaxel regimens.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* breast cancer stages II-III
* adjuvant or neoadjuvant chemotherapy with docetaxel regimens (TAC or anthracyclines followed by docetaxel 100 mg/m2 x 4)

Exclusion Criteria:

* contraindications for adjuvant docetaxel and or anthracyclines

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
percentage of patients without persistent alopecia | 2nd year following docetaxel chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: miguel martin, MD, PHD, Principal Investigator — hospital clinico san carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Martin M, de la Torre-Montero JC, Lopez-Tarruella S, Pinilla K, Casado A, Fernandez S, Jerez Y, Puente J, Palomero I, Gonzalez Del Val R, Del Monte-Millan M, Massarrah T, Vila C, Garcia-Paredes B, Garcia-Saenz JA, Lluch A. Persistent major alopecia following adjuvant docetaxel for breast cancer: incidence, characteristics, and prevention with scalp cooling. Breast Cancer Res Treat. 2018 Oct;171(3):627-634. doi: 10.1007/s10549-018-4855-2. Epub 2018 Jun 19. PMID 29923063